CLINICAL TRIAL: NCT03822507
Title: A Phase 3, Randomized, Double-Blind, Intra-Subject Dose-Adjustment, Parallel-Group Study of KHK7580 and Cinacalcet Hydrochloride in Subjects With Secondary Hyperparathyroidism Receiving Hemodialysis
Brief Title: Study of KHK7580 in Subjects With Secondary Hyperparathyroidism in Asia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Kirin China Pharmaceutical Co., Ltd. (Industry); Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7580-201
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHK7580 1mg-12mg (Experimental)
  Interventions: Drug: KHK7580
- Cinacalcet 25mg-100mg (Active Comparator)
  Interventions: Drug: Cinacalcet Hydrochloride

INTERVENTIONS:
Drug: KHK7580 — oral administration
  Arms: KHK7580 1mg-12mg
Drug: Cinacalcet Hydrochloride — oral administration
  Arms: Cinacalcet 25mg-100mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of KHK7580 orally administered once daily for 52 weeks compared to cinacalcet hydrochloride as an active control in subjects with secondary hyperparathyroidism receiving hemodialysis in China, Korea, Hong Kong and Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Personally submitted written voluntary informed consent to participate in the study
2. Aged ≧18 years at the time of consent
3. Stable chronic renal failure treated with hemodialysis 3 times weekly for at least 12 weeks before screening
4. Intact PTH level (centrally measured) of >300 pg/mL at screening
5. Corrected serum Ca level (centrally measured) of ≧9.0 mg/dL at screening

Exclusion Criteria:

1. Treatment with cinacalcet hydrochloride within 2 weeks before screening
2. Change in dose or dosing regimen of an activated vitamin D drug or its derivative, phosphate binder, or Ca preparation within 2 weeks before screening; or start of treatment with such drugs within 2 weeks before screening
3. Change in prescribed conditions of dialysis (dialysate Ca concentration, prescribed dialysis time, and prescribed number of dialysis per week) within 2 weeks before screening
4. Treatment with bisphosphonates, denosumab or teriparatide within 24 weeks before screening
5. Parathyroidectomy and/or parathyroid intervention within 24 weeks before screening
6. Severe heart disease (e.g., ≧ Class Ⅲ per New York Heart Association classification)
7. Severe hepatic dysfunction (e.g., treatment with antiviral therapy)
8. Uncontrolled hypertension and/or diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Mean percent change in intact parathyroid hormone (PTH) level from baseline in the evaluation period | Week 50- Week 52

SECONDARY OUTCOMES:
Number of subjects achieving a mean intact PTH level of ≧150pg/mL and ≦300pg/mL in the evaluation period | Week 50- Week 52
Percentage of subjects achieving a mean intact PTH level of ≧150pg/mL and ≦300pg/mL in the evaluation period | Week 50- Week 52
Number of subjects achieving a mean percent decrease in intact PTH level of ≧３０% (percent change ≦-３０%) from baseline in the evaluation period | Week 50- Week 52
Percentage of subjects achieving a mean percent decrease in intact PTH level of ≧３０% (percent change ≦-３０%) from baseline in the evaluation period | Week 50- Week 52
Intact PTH level | Week 50- Week 52
corrected serum Ca level | Week 50- Week 52
serum P level | Week 50- Week 52

CONTACTS AND LOCATIONS:
Locations (34):
- China (13):
  - Research site_29, Changsha
  - Research site_34, Dalian
  - Research site_25, Foshan
  - Research site_22, Guangzhou
  - Research site_23, Guangzhou
  - Research site_30, Guangzhou
  - Research site_28, Hefei
  - Research site_32, Nanjing
  - Research site_33, Nanjing
  - Research site_24, Shanghai
  - Research site_26, Shanghai
  - Research site_27, Shanghai
  - Research site_31, Wuxi
- Research site_11, Hong Kong, Hong Kong
- South Korea (10):
  - Research site_21, Anyang
  - Research site_13, Daegu
  - Research site_15, Daegu
  - Research site_12, Goyang
  - Research site_18, Incheon
  - Research site_14, Seoul
  - Research site_17, Seoul
  - Research site_19, Seoul
  - Research site_20, Seoul
  - Research site_16, Ulsan
- Taiwan (10):
  - Research site_2, Kaohsiung City
  - Research site_3, Kaohsiung City
  - Research site_5, Kaohsiung City
  - Research site_9, Taichung
  - Research site_4, Tainan
  - Research site_7, Tainan
  - Research site_10, Taipei
  - Research site_1, Taipei
  - Research site_6, Taipei
  - Research site_8, Taipei

IPD SHARING:
Plan to Share IPD: No